CLINICAL TRIAL: NCT05545163
Title: Comparison of Simulated Standard Versus Modified Jaw Thrust I-gel Insertion Technique in Novice Anesthesiologists: A Randomised Control Crossover Trial
Brief Title: Comparison of Simulated Standard Versus Modified Jaw Thrust I-gel Insertion Technique in Novice Anesthesiologists
Acronym: I-gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dileep Kumar, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2021-6257-21893
Record Dates: First submitted 2022-09-13; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Training Group, Sensitivity; Igel
Keywords: I-gel; Technique; Standard; Modified; Simulation
MeSH Terms: conditions — Hypersensitivity; Ige Responsiveness, Atopic

STUDY DESIGN:
Intervention Model Description: Each novice resident will place ten times I-gel insertion with each insertion technique in randomized cross over manner by dividing the residents in two groups (5 residents in each group), by draw method. The one group will place I-gel with standard insertion technique and other group will place by modified jaw thrust I-gel insertion technique, then after, the groups will switch over with concerned insertion techniques
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-gel with standard insertion technique (No Intervention): in this arm, trainees performed the standard I-gel insertion technique
- Modified jaw thrust I-gel insertion technique (Experimental): in this arm, trainees performed modified jaw thrust insertion technique
  Interventions: Device: I-gel with standard insertion technique

INTERVENTIONS:
Device: I-gel with standard insertion technique — Standard I-gel insertion technique (grasping I-gel from integral bite block site and cuff facing towards chin and pressing down the manikin chin. I-gel introduced in patient's mouth in a direction towards hard palate. Then I-gel slided downwards and backwards along hard palate with a continuous but gentle push until a definitive resistance is felt)
  Modified jaw thrust technique (grasping I-gel from integral bite block site and cuff facing towards chin and pressing down manikin chin. I-gel introduced in patient's mouth in a direction towards hard palate with gently advancing into oropharynx. Then after, I-gel left in oral cavity and both hands used to thrust jaw by lifting angle of mandible with little fingers and other fingers to stabilise jaw. And, at this point, both hand's thumbs used to apply balance force from I-gel stem head towards final placement position by looking at integral bite block mark at incisor teeth level)
  Other Names: Modified jaw thrust I-gel insertion technique
  Arms: Modified jaw thrust I-gel insertion technique

SUMMARY:
The primary objective of study was to compare insertion ease by modified I-gel jaw thrust insertion technique and standard I-gel insertion technique on the basis of I-gel insertion attempts and I-gel insertion time duration. The secondary objective of study was to analyse the impact of prior information for airway device, insertion techniques, general or specific work experience in airway management with the ease of both study's insertion techniques. And, tertiary objective of study was to analyse the trainee's preference insertion technique at the basis of learning method and practical adaptability.

Hypothesis:

The modified I-gel jaw thrust insertion technique is easy to understand and practice than the standard I-gel insertion technique at the beginning of airway management training among the novice anesthesiologists.

DETAILED DESCRIPTION:
* I-gel insertion attempts are the number of I-gel insertion attempts with each study's insertion technique. The 10 insertion attempts allowed to performed with each insertion technique by trainees.
* I-gel insertion time duration was the time taken to complete I-gel insertion; from the holding of device till the confirmation of chest movement (artificial lung inflation in manikin).
* The correlation of previous information for airway device, insertion techniques, general or specific work experience in airway management with the ease of both study's insertion techniques were assessed by asking from participant's questionnaire based at the start of study.
* The trainees were asked at the end of study for preferred insertion method at novice level on the basis of learning method and practical conduct (user friendly).

ELIGIBILITY:
Inclusion Criteria:

* First year anaesthesia residents
* Using adult mannequin

Exclusion Criteria:

* Pediatric mannequin
* Participant's refusal

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2021-10-02 (Actual); Study Completion 2021-10-02 (Actual)

PRIMARY OUTCOMES:
The ease of I-gel insertion was measured on the basis of number of I-gel insertion attempts. | 5 minutes
  Ease of I-gel insertion in mannequin mouth was measured by performing the 10 times insertion of I-gel with both study techniques in mannequin mouth by trainees.
The ease of I-gel insertion was measured on the basis of final I-gel insertion time taken duration. | 5 minutes
  The total time duration of final I-gel insertion confirmation in mannequin mouth was recorded. The time duration counting was started from I-gel holding in operator's hand to the confirmed successful insertion in mannequin mouth.

SECONDARY OUTCOMES:
The trainee's baseline knowledge was assessed for the type of supraglottic airway devices and I-gel insertion techniques. | 1 minute
  The questionnaire based trainee's asked for the prior information of the I-gel and other supraglottic airway device.
The trainee's baseline knowledge was assessed for the type I-gel insertion techniques. | 1 minute
  The questionnaire based trainee's asked for the prior information for the type of I-gel insertion techniques.
The trainee's baseline knowledge was assessed for the general or specific work experience in airway management using the I-gel. | 1 minute
  The questionnaire based trainee's asked for previous experience in using the I-gel device.
The trainee's baseline knowledge was assessed for the studied modified jaw thrust I-gel insertion technique. | 2 minutes
  The questionnaire based trainee's asked for the previous experience for modified jaw thrust I-gel insertion technique.

OTHER OUTCOMES:
The trainee's asked for the choice of I-gel insertion technique at the start of learning airway management using the I-gel at his level | 2 minutes
  The questionnaire based trainee's asked for the choice of type of I-gel insertion technique such as standard or modified jaw thrust insertion at start of learning the airway management at his level of training year.
The trainee's asked for the easy learning of I-gel insertion technique at his level of training. | 2 minutes
  The questionnaire based trainee's asked for his experience of easy learning of type of I-gel insertion technique such as standard or modified jaw thrust insertion at his level of training year.
The trainee's asked for the preference of I-gel insertion technique in his practice at his level of training. | 1 minute
  The questionnaire based trainee's asked for his preference to practice most of the time for the type of I-gel insertion technique like standard or modified jaw thrust insertion at his level of training year.

CONTACTS AND LOCATIONS:
Overall Officials: dileep kumar, MD, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the study and consent has been taken from participants.
Supporting Information: SAP, CSR
Time Frame: Data is available
Access Criteria: Through Publication only
URL: https://www.aku.edu

REFERENCES:
- [Background] Boet S, Borges BC, Naik VN, Siu LW, Riem N, Chandra D, Bould MD, Joo HS. Complex procedural skills are retained for a minimum of 1 yr after a single high-fidelity simulation training session. Br J Anaesth. 2011 Oct;107(4):533-9. doi: 10.1093/bja/aer160. Epub 2011 Jun 9. PMID 21659406
- [Background] Kennedy CC, Cannon EK, Warner DO, Cook DA. Advanced airway management simulation training in medical education: a systematic review and meta-analysis. Crit Care Med. 2014 Jan;42(1):169-78. doi: 10.1097/CCM.0b013e31829a721f. PMID 24220691
- [Background] Sun Y, Pan C, Li T, Gan TJ. Airway management education: simulation based training versus non-simulation based training-A systematic review and meta-analyses. BMC Anesthesiol. 2017 Feb 1;17(1):17. doi: 10.1186/s12871-017-0313-7. PMID 28143389
- [Background] Lee DW, Kang MJ, Kim YH, Lee JH, Cho KW, Kim YW, Cho JH, Kim YS, Hong CK, Hwang SY. Performance of intubation with 4 different airway devices by unskilled rescuers: manikin study. Am J Emerg Med. 2015 May;33(5):691-6. doi: 10.1016/j.ajem.2015.03.006. Epub 2015 Mar 12. PMID 25800412
- [Background] Jackson KM, Cook TM. Evaluation of four airway training manikins as patient simulators for the insertion of eight types of supraglottic airway devices. Anaesthesia. 2007 Apr;62(4):388-93. doi: 10.1111/j.1365-2044.2007.04983.x. PMID 17381577
- [Background] Kumar D, Hayat M, Khan A. i-gel insertion with modified jaw thrust technique. Indian J Anaesth. 2015 Feb;59(2):132-3. doi: 10.4103/0019-5049.151383. No abstract available. PMID 25788752
- [Background] Bhardwaj M, Singhal SK, Rashmi, Dahiya A. A prospective randomised trial to compare three insertion techniques for i-gel placement: Standard, reverse, and rotation. Indian J Anaesth. 2020 Jul;64(7):618-623. doi: 10.4103/ija.IJA_937_19. Epub 2020 Jul 1. PMID 32792739